CLINICAL TRIAL: NCT06965764
Title: Study of Contrast - Induced Nephropathy After Intravenous Contrast Procedures at Sohag University Hospitals
Status: Recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Esraa Ragab Youssef, Principal Investigator, Internal Medicine Resident, Sohag University
Other Study IDs: Soh-Med--25-3-03MS
Record Dates: First submitted 2025-04-16; First posted 2025-05-11 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-03

CONDITIONS: Contract Induced Nephropathy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Contrast-induced nephropathy (CIN) is a serious complication of angiographic procedures and results from administration of iodinated contrast media (CM).

CIN is the third most common cause of hospital acquired acute renal injury representing about 12% of the cases. The reported incidence of CIN varies widely across the literature, depending on the patient population studied and the baseline risk factors . An overall incidence of CIN following intraarterial contrast injection in the general population was reported to be 0.6-2.3%.

Although the incidence of CIN is low in patients with normal renal function, its prevalence can be much higher in several patient subsets e.g. diabetics, patients with existing renal insufficiency.

Contrast-induced nephropathy is defined as a rise in serum creatinine of at least 0.5 mg/dL or a 25% increase from baseline within 48 to 72 hours after contrast exposure. The Kidney Disease Improving Global Outcome (KDIGO) definition is different, with stage 1 being a rapid rise of creatinine to greater than 0.3 mg/dL within 48 hours or the relative rise of 50% or more from baseline in 7 days or less or a reduction in urine output to less than 0.5 ml/kg/hr for 6 to 12 hours. This severity is further staged based on creatinine levels, urine output, or the need for renal replacement therapy.

In most cases of CIN there is an asymptomatic, non-oliguric rise of serum creatinine within 24hours; however, in more severe cases, the creatinine concentration may not peak until 5-10 days and the increase may be associated with oliguria, It may occasionally progress to end-stage renal failure.

The incidence of CIN varies widely among the publications in the literature and studies. In this study, we will evaluate the incidence of CIN amongst patients receiving intravenous contrast in sohag university hospital, to study the variations in serum creatinine levels with contrast administration.

ELIGIBILITY:
Inclusion Criteria:

1- Inpatients and outpatients aged 18years and above who underwent single intravenous Contrast procedures.

Exclusion criteria:

1. Patients below 18 years, failure to obtain consent.
2. Patients with ESRD/ on maintenance hemodialysis.
3. New-York Heart Association class IV Congestive Cardiac Failure (CCF) or patients with cardiogenic shock .
4. History of hypersensitivity to contrast in the past or exposure to contrast in the last 24-48 hours, 5-nursing/pregnant subjects.
5. Patients with malignancy or other organ failure like decompensated liver cirrhosis

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inpatients and outpatients aged 18years and above who underwent single intravenous Contrast procedures
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-03-12 (Actual); Primary Completion 2025-09-12 (Estimated); Study Completion 2025-09-12 (Estimated)

PRIMARY OUTCOMES:
Title: Incidence of Contrast-Induced Nephropathy (CIN) | Within 48-72 hours after contrast administration
  increase in serum creatinine by ≥0.5 mg/dL or ≥25% from baseline. Serum creatinine will be measured before and 48-72 hours after contrast exposure.

SECONDARY OUTCOMES:
Correlation between Risk Factors and Development of Contrast-Induced Nephropathy (CIN) | At the time of enrollment and after 72 hours of contrast exposure
  This outcome assesses the correlation between the presence of risk factors - including age (in years), diabetes mellitus (yes/no), and baseline renal function [estimated GFR in mL/min/1.73m², measured using the CKD-EPI equation] - and the incidence of Contrast-Induced Nephropathy (CIN), defined as an increase in serum creatinine by ≥0.5 mg/dL or ≥25% from baseline.
  CIN will be assessed within 48-72 hours after contrast administration. The correlation will be measured using multivariate logistic regression analysis or Spearman's correlation as appropriate.

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university hospitals, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided